CLINICAL TRIAL: NCT01145105
Title: Efficacy of Neural Dynamics Technique in the Treatment of Chronic Low Back Pain With Radiation to the Leg
Brief Title: Neural Dynamics Technique for the Treatment of Chronic Radicular Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Uzi Milman, Uzi Milman MD, Clinical Research Unit, Clalit Health Services, Haifa District, HAIFA, ISRAEL., Clalit Health Services
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-09-0078-ctil
Record Dates: First submitted 2010-05-24; First posted 2010-06-16 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-07

CONDITIONS: Low Back Pain; Sciatica
Keywords: Low back pain; Sciatica; Pain; Physiotherapy
MeSH Terms: conditions — Low Back Pain; Sciatica; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: neural dynamics techniques treatment — Treatment group- will receive neural mobilizations techniques, to improve movement of the sciatic nerve.
  Other Names: Physiotherapy
Procedure: placebo treatment — Control group- will receive placebo treatment that will include mobilization to the upper limb. After the placebo treatment, these patients will receive neural mobilizations techniques.
  Other Names: physiotherapy

SUMMARY:
Low back pain ( LBP) is a significant health problem which affects about 70%-80% of the population during the course of their life . The majority of LBP is resolved within 3 months; however, up to 40% of LBP becomes chronic. One subgroup of chronic LBP is patients with sciatica. Sciatica is characterized by radiating pain to the buttock and lower limb, with or without low back pain.

It has been shown in the upper limb that by positioning the contra-lateral arm in tension the investigators actually reduce tension in the ipsilateral arm. Patients, who present with symptoms like sciatica, can benefit from this maneuver (neural dynamics techniques) that reduces tension through the contra-lateral leg.

Working Hypothesis: Compared with a placebo maneuver of the upper limb, the neural dynamics techniques will result in better rehabilitation of individuals with radicular LBP.

DETAILED DESCRIPTION:
Objectives: To evaluate the efficacy of neural dynamics techniques, using the contra-lateral leg, in the treatment of sub-acute/chronic Low back pain with radiation to the leg. Study Methodology: Eligible individuals will be assessed by a physiotherapist that will be blinded to the treatment allocation; treatment (either intervention or placebo) will be provided by a physiotherapist that will be blinded to the patient's assessment. The treated individuals and the referring physician will also be blinded to the treatment allocation;

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* LBP with radiation to one leg, that lasts more than 6 weeks
* Abnormal response to SLR test
* With or without neurological signs

Exclusion Criteria:

* History of spinal surgery
* Patient with FUO
* History of malignancies
* Patient with saddle anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of neural dynamics technique | 5 weeks
  Efficacy will be measured by combining 5 tools
  1. Oswestry disability index.
  2. McGill Pain Questionnaire
  3. Visual analog scale for pain assessment.
  4. Lumbar flexion measurement (the distance of the tip of the index finger to the inferior angle of the Patella, measured by a measurement tape.
  5. Passive SLR range of motion- measured with inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Noga Roguin Maor, MD, Principal Investigator — clinical research unit, Clalit health services, Haifa and western Galilee district.; Uzi Milman, MD, Study Director — clinical research unit, Clalit health services, Haifa and western Galilee district.
Locations (1):
- Clalit Health Services, Haifa and Western Galilee District, Haifa, Israel